CLINICAL TRIAL: NCT06158152
Title: A Randomized, Double-blind, Placebo-controlled Pilot Study to Evaluate the Systemic Effect on Immunoinflammatory and Metabolic Status of an Oral Supplementation With AM3 in Patients With Metabolic Syndrome.
Brief Title: A Pilot Study to Evaluate the Systemic Effect of Oral Supplementation With AM3 in Patients With Metabolic Syndrome.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Industrial Farmacéutica Cantabria, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: P20110a
Record Dates: First submitted 2023-07-26; First posted 2023-12-06 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic Syndrome; AM3; Probiotics; Inmunoferon; Food suplement; Immune response
MeSH Terms: conditions — Metabolic Syndrome | interventions — Immunoferon; Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Active arm (Active Comparator): Patients who will receive the study treatment (AM3 Technology in combination with Probiotic SynBalance Metsyn)
  Interventions: Dietary Supplement: AM3 + Probiotic
- Placebo arm (Placebo Comparator): Patients who will receive placebo treatment, consisting of starch capsules
  Interventions: Dietary Supplement: Placebo
- Control arm (Sham Comparator): Patients to be treated with AM3 Technology capsules
  Interventions: Dietary Supplement: AM3

INTERVENTIONS:
Dietary Supplement: AM3 + Probiotic — Two capsules daily in the morning during 12 weeks. The capsule contains the mixture of AM3 Technology and probiotic SynBalance Metsyn.
  Arms: Active arm
Dietary Supplement: Placebo — Two capsules daily in the morning during 12 weeks. The capsule contains starch.
  Arms: Placebo arm
Dietary Supplement: AM3 — Two capsules daily in the morning during 12 weeks. The capsule contains AM3 Technology.
  Arms: Control arm

SUMMARY:
The goal of this pilot study is to learn about the effect of the nutritional supplementation based on AM3 in combination with probiotics on imflammatory and metabolic mediators in adult subjects diagnosed with metabolic syndrome.

The hypothesis the investigators are testing focuses on the fact that the continued use of the nutritional supplement with AM3 and probiotics is capable of minimizing the risk factors associated with metabolic syndrome, by reducing the development of the derived chronic pathologies.

A total of 48 subjects with a diagnosis of metabolic syndrome is planned to be recruited from two investigational sites in the Comunity of Madrid (Spain). These subjects will be randomized into three treatment groups (active, placebo, and control). The dosage will be of 2 capsules/day in a single intake in the morning for 12 weeks. Two interventional visits are planned to be performed: at baseline and at week 12.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, pilot study. The primay objective is to evaluate the systemic effect of this new nutritional supplement with AM3 and probiotics on the immuno-inflammatory and metabolic status against metabolic syndrome.

The secondary objectives are:

1. To determine the efficacy of the administration of a new food supplement for MS through the improvement of biochemical variables.
2. To evaluate the efficacy of the administration of a new dietary supplement on the impact on body composition parameters.
3. To evaluate the patient's quality of life.

Adult subjects (aged between 18 and 75 years) will randomly be assigned into one of these three treatment groups:

* Active: patients who will receive the study treatment, consisting of the combination of AM3 and the probiotic SynBalance Metsyn.
* Placebo: patients who will receive placebo (starch capsules), with no active ingredient.
* Control: patients to be treated with AM3 capsules alone (no probiotics).

Interventions performed at time 0 and 12 weeks, are carried out to measure parameters such as the following: body composition data (weight, BMI), blood pressure, fasting glucose and insulin levels, monocyte and NK-cell populations, liver enzyme levels, urine sediment, etc.

Finally, a subjective questionnaire is used to evaluate the patients' quality of life before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged 18-75 years at the time of signing the informed consent form.
2. Diagnosis of metabolic syndrome, defined as: central obesity, elevation of blood glucose by ≥100 mg/dl, glycosylated hemoglobin between 5.7 and 6.4%, low HDL cholesterol levels < 40 mg/dl in men and < 50 mg/dl in women, and high levels of triglycerides, being higher than 150 mg/dl.
3. If the patient is being treated with metformin, lipid-lowering treatment with statins or treatment with antihypertensives, he/she must have a stable dose at the time of inclusion.

Exclusion Criteria:

1. Smokers or with history of alcoholism or drug abuse .
2. To have hypertriglyceridemia (> 500 mg/dL).
3. Uncontrolled arterial hypertension, as per investigator's criteria.
4. To have undergone bariatric surgery over the last 24 months that according to investigator's criteria, this might interfere with his/her participation in the study.
5. Diagnosis of chronic diseases that according to investigator's criteria, this might interfere with his/her participation in the study.
6. Presence of renal insufficiency (glomerular filtration rate below 30 ml/minute).
7. Presence of severe respiratory insufficiency (PaO2 less than 60 mmHg or PaCO2 greater than 50 mmHg).
8. Presence of heart failure (LVEF <30% and RVEF <35%).
9. Presence of the following diseases in an unstable manner, according to the investigator's criteria: chronic obstructive disease, inflammatory bowel disease, intestinal malabsorption syndrome, systemic autoimmune diseases, rheumatoid arthritis, spondyloarthritis, psoriasis, and chronic inflammatory skin diseases.
10. Active or chronic severe unstable infections that, in medical criteria, may interfere with patients' safety.
11. Disease-related malnutrition.
12. Endocrinologic unestable or uncontrolled diseases that in medical criteria, present with manifestations in pituitary, adrenal or thyroid function.
13. Immunosuppressive or corticosteroid treatment in the last 3 months.
14. Treatment with semaglutide and tirzepatide.
15. Pregnant women (or intending to become pregnant) or breast-feeding women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in serum cytokines. | Baseline and week 12
  Circulating cytokine levels will be determined at baseline and at week 12 to assess the effect on inflammatory mediators.

SECONDARY OUTCOMES:
Change in monocytes and natural killer cells levels. | Baseline and week 12
  Serum monocytes and natural killers cells will be determined at baseline and week 12 to assess the effect on inflammatory status and oxidative stress.
Change in serum uric acid. | Baseline and week 12
  Uric acid will be analized to assess the effect on inflammatory and metabolic mediators. These results will be displayed in the results data table.
Change in serum sodium. | Baseline and week 12
  sodium will be analized to assess the effect on inflammatory and metabolic mediators. These results will be displayed in the results data table.
Change in serum potasium. | Baseline and week 12
  potassium will be analized to assess the effect on inflammatory and metabolic mediators. These results will be displayed in the results data table.
Change in serum bilirrubin. | Baseline and week 12
  Bilirrubin will be analized to assess the effect on inflammatory and metabolic mediators. These results will be displayed in the results data table.
Change in serum lipids | Baseline and week 12
  Serum lipids will be determined at baseline and at week 12 to assess the effect on metabolic parameters.
Change in serum glucose | Baseline and week 12
  Fasting blood glucose levels will be analized to assess the effect on inflammatory and metabolic mediators.
Change in blood pressure | Baseline and week 12.
  Blood pressure (Diastolic and systolic) [mmHg] will be determined at baseline and after 12 weeks of study treatment.
Change in waist circumference | Baseline and week 12
  Waist circumference [cm] will be obtained at baseline and at week 12 to assess the efficacy on body composition.
Change in hip circumference | Baseline and week 12
  Hip circumference [cm] will be obtained at baseline and at week 12 to assess the efficacy on body composition.
Change in weight | Baseline and week 12
  Weight [Kg] will be obtained at baseline and at week 12 to assess the efficacy on body composition. These results will be displayed in the results data table.
Change in body mass index | Baseline and week 12
  BMI [Kg/m2] will be obtained at baseline and at week 12 to assess the efficacy on body composition. These results will be displayed in the results data table.
Change in total body fat content | Baseline and week 12
  Total body fat content will be measured at baseline and at week 12 using electrical bioimpedance.
Change in patient's quality of life, assessed by the SF-12v2 score. | Baseline and week 12
  This is a health-related quality-of-life questionnaire, consisting of 12 questions that measure eight health domains to assess physical and mental health. Physical health-related domains include General Health (GH), Physical Functioning (PF), Role Physical (RP), and Body Pain (BP). This score will be determined at baseline and at week 12.
  Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Álvarez, Principal Investigator — Servicio de Endocrinología y Nutrición del Hospital Universitario Príncipe de Asturias de Alcalá de Henares (Madrid)
Locations (2):
- Spain (2):
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario Príncipe de Asturias, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Francisco V, Ruiz-Fernandez C, Pino J, Mera A, Gonzalez-Gay MA, Gomez R, Lago F, Mobasheri A, Gualillo O. Adipokines: Linking metabolic syndrome, the immune system, and arthritic diseases. Biochem Pharmacol. 2019 Jul;165:196-206. doi: 10.1016/j.bcp.2019.03.030. Epub 2019 Mar 22. PMID 30910694
- [Background] Mendrick DL, Diehl AM, Topor LS, Dietert RR, Will Y, La Merrill MA, Bouret S, Varma V, Hastings KL, Schug TT, Emeigh Hart SG, Burleson FG. Metabolic Syndrome and Associated Diseases: From the Bench to the Clinic. Toxicol Sci. 2018 Mar 1;162(1):36-42. doi: 10.1093/toxsci/kfx233. PMID 29106690
- [Background] Grandl G, Wolfrum C. Hemostasis, endothelial stress, inflammation, and the metabolic syndrome. Semin Immunopathol. 2018 Feb;40(2):215-224. doi: 10.1007/s00281-017-0666-5. Epub 2017 Dec 5. PMID 29209827
- [Background] Wang Q, Wu H. T Cells in Adipose Tissue: Critical Players in Immunometabolism. Front Immunol. 2018 Oct 30;9:2509. doi: 10.3389/fimmu.2018.02509. eCollection 2018. PMID 30459770
- [Background] Guerrero A, Brieva A, Pivel JP. A new method for radioiodination of polysaccharides and its use in biodistribution studies of an immunomodulating glycoconjugate (Immunoferon). Methods Find Exp Clin Pharmacol. 2000 Oct;22(8):621-5. doi: 10.1358/mf.2000.22.8.802273. PMID 11256233
- [Background] Vega-Robledo GB, Rico-Rosillo MG. [Adipose tissue: immune function and alterations caused by obesity]. Rev Alerg Mex. 2019 Jul-Sep;66(3):340-353. doi: 10.29262/ram.v66i3.589. Spanish. PMID 31606018
- [Background] Varela J, Navarro Pico ML, Guerrero A, Garcia F, Gimenez Gallego G, Pivel JP. Identification and characterization of the peptidic component of the immunomodulatory glycoconjugate Immunoferon. Methods Find Exp Clin Pharmacol. 2002 Oct;24(8):471-80. doi: 10.1358/mf.2002.24.8.705066. PMID 12500425
- [Background] Ortega del Alamo P, Rivera Rodriguez T, Sanz Fernandez R. [The effect of AM3 in the resolution of otitis media with effusion (OME) in paediatric patients]. Acta Otorrinolaringol Esp. 2005 Jan;56(1):1-5. doi: 10.1016/s0001-6519(05)78561-7. Spanish. PMID 15747716
- [Background] King GL. The role of inflammatory cytokines in diabetes and its complications. J Periodontol. 2008 Aug;79(8 Suppl):1527-34. doi: 10.1902/jop.2008.080246. PMID 18673007
- [Background] Donath MY, Dinarello CA, Mandrup-Poulsen T. Targeting innate immune mediators in type 1 and type 2 diabetes. Nat Rev Immunol. 2019 Dec;19(12):734-746. doi: 10.1038/s41577-019-0213-9. Epub 2019 Sep 9. PMID 31501536
- [Background] Remely M, Hippe B, Zanner J, Aumueller E, Brath H, Haslberger AG. Gut Microbiota of Obese, Type 2 Diabetic Individuals is Enriched in Faecalibacterium prausnitzii, Akkermansia muciniphila and Peptostreptococcus anaerobius after Weight Loss. Endocr Metab Immune Disord Drug Targets. 2016;16(2):99-106. doi: 10.2174/1871530316666160831093813. PMID 27577947
- [Background] Serrano-Gomez D, Martinez-Nunez RT, Sierra-Filardi E, Izquierdo N, Colmenares M, Pla J, Rivas L, Martinez-Picado J, Jimenez-Barbero J, Alonso-Lebrero JL, Gonzalez S, Corbi AL. AM3 modulates dendritic cell pathogen recognition capabilities by targeting DC-SIGN. Antimicrob Agents Chemother. 2007 Jul;51(7):2313-23. doi: 10.1128/AAC.01289-06. Epub 2007 Apr 23. PMID 17452477
- [Background] Prieto A, Reyes E, Bernstein ED, Martinez B, Monserrat J, Izquierdo JL, Callol L, de LUCAS P, Alvarez-Sala R, Alvarez-Sala JL, Villarrubia VG, Alvarez-Mon M. Defective natural killer and phagocytic activities in chronic obstructive pulmonary disease are restored by glycophosphopeptical (inmunoferon). Am J Respir Crit Care Med. 2001 Jun;163(7):1578-83. doi: 10.1164/ajrccm.163.7.2002015. PMID 11401877
- [Background] Brieva A, Guerrero A, Alonso-Lebrero JL, Pivel JP. Immunoferon, a glycoconjugate of natural origin, inhibits LPS-induced TNF-alpha production and inflammatory responses. Int Immunopharmacol. 2001 Oct;1(11):1979-87. doi: 10.1016/s1567-5769(01)00125-4. PMID 11606029
- [Background] Majano P, Alonso-Lebrero JL, Janczyk A, Martin-Vichez S, Molina-Jimenez F, Brieva A, Pivel JP, Gonzalez S, Lopez-Cabrera M, Moreno-Otero R. AM3 inhibits LPS-induced iNOS expression in mice. Int Immunopharmacol. 2005 Jul;5(7-8):1165-70. doi: 10.1016/j.intimp.2005.02.009. Epub 2005 Mar 16. PMID 15914321
- [Background] Hills RD Jr, Pontefract BA, Mishcon HR, Black CA, Sutton SC, Theberge CR. Gut Microbiome: Profound Implications for Diet and Disease. Nutrients. 2019 Jul 16;11(7):1613. doi: 10.3390/nu11071613. PMID 31315227
- [Background] Cicero AFG, Fogacci F, Bove M, Giovannini M, Borghi C. Impact of a short-term synbiotic supplementation on metabolic syndrome and systemic inflammation in elderly patients: a randomized placebo-controlled clinical trial. Eur J Nutr. 2021 Mar;60(2):655-663. doi: 10.1007/s00394-020-02271-8. Epub 2020 May 16. PMID 32417946
- [Background] Borchers A, Pieler T. Programming pluripotent precursor cells derived from Xenopus embryos to generate specific tissues and organs. Genes (Basel). 2010 Nov 18;1(3):413-26. doi: 10.3390/genes1030413. PMID 24710095
- [Background] Monserrat J, Asunsolo A, Gomez-Lahoz A, Ortega MA, Gasalla JM, Gasulla O, Fortuny-Profitos J, Mazaira-Font FA, Teixido Roman M, Arranz A, Sanz J, Munoz B, Arevalo-Serrano J, Rodriguez JM, Martinez-A C, Balomenos D, Alvarez-Mon M. Impact of the Innate Inflammatory Response on ICU Admission and Death in Hospitalized Patients with COVID-19. Biomedicines. 2021 Nov 12;9(11):1675. doi: 10.3390/biomedicines9111675. PMID 34829906
- [Background] Alvarez-Mon MA, Ortega MA, Garcia-Montero C, Fraile-Martinez O, Lahera G, Monserrat J, Gomez-Lahoz AM, Molero P, Gutierrez-Rojas L, Rodriguez-Jimenez R, Quintero J, Alvarez-Mon M. Differential malondialdehyde (MDA) detection in plasma samples of patients with major depressive disorder (MDD): A potential biomarker. J Int Med Res. 2022 May;50(5):3000605221094995. doi: 10.1177/03000605221094995. PMID 35615790
- [Background] Alvarez-Mon M, Ortega MA, Gasulla O, Fortuny-Profitos J, Mazaira-Font FA, Saurina P, Monserrat J, Plana MN, Troncoso D, Moreno JS, Munoz B, Arranz A, Varona JF, Lopez-Escobar A, Barco AA. A Predictive Model and Risk Factors for Case Fatality of COVID-19. J Pers Med. 2021 Jan 8;11(1):36. doi: 10.3390/jpm11010036. PMID 33430129
- [Background] Ortega MA, Fraile-Martinez O, Garcia-Montero C, Alvarez-Mon MA, Gomez-Lahoz AM, Albillos A, Lahera G, Quintero J, Monserrat J, Guijarro LG, Alvarez-Mon M. An Updated View of the Importance of Vesicular Trafficking and Transport and Their Role in Immune-Mediated Diseases: Potential Therapeutic Interventions. Membranes (Basel). 2022 May 25;12(6):552. doi: 10.3390/membranes12060552. PMID 35736259
- [Background] Lario M, Munoz L, Ubeda M, Borrero MJ, Martinez J, Monserrat J, Diaz D, Alvarez-Mon M, Albillos A. Defective thymopoiesis and poor peripheral homeostatic replenishment of T-helper cells cause T-cell lymphopenia in cirrhosis. J Hepatol. 2013 Oct;59(4):723-30. doi: 10.1016/j.jhep.2013.05.042. Epub 2013 Jun 3. PMID 23742913
- [Background] Albillos A, de la Hera A, Gonzalez M, Moya JL, Calleja JL, Monserrat J, Ruiz-del-Arbol L, Alvarez-Mon M. Increased lipopolysaccharide binding protein in cirrhotic patients with marked immune and hemodynamic derangement. Hepatology. 2003 Jan;37(1):208-17. doi: 10.1053/jhep.2003.50038. PMID 12500206
- [Background] Alvarez-Mon MA, Gomez-Lahoz AM, Orozco A, Lahera G, Diaz D, Ortega MA, Albillos A, Quintero J, Auba E, Monserrat J, Alvarez-Mon M. Expansion of CD4 T Lymphocytes Expressing Interleukin 17 and Tumor Necrosis Factor in Patients with Major Depressive Disorder. J Pers Med. 2021 Mar 19;11(3):220. doi: 10.3390/jpm11030220. PMID 33808804
- See also: Inflammation and insulin resistance: mechanisms for the endothelial dysfunction development and atherosclerosis. — https://www.medigraphic.com/pdfs/cardio/h-2006/h062a.pdf
- See also: Immunopathogenesis of aging: the impairment of innate immunity and its impact on specific immunity. Restoration by AM3. — https://www.elsevier.es/es-revista-revista-espanola-geriatria-gerontologia-124-pdf-13006144